CLINICAL TRIAL: NCT03839914
Title: Randomized, Controlled, Single-blinded Trial to Evaluate the Efficacy and Safety of Intra-wound Administration of Vancomycin Powder as Add-on Prophylactic Intraoperative Antibiotic in Patients at High Risk for Surgical Site Infections After Receiving Open Posterior Spinal Surgery
Brief Title: Evaluating the Efficacy and Safety of Intra-wound Vancomycin Powder in High Risk Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Jason Pui Yin Cheung, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Study protocol 1.4
Record Dates: First submitted 2019-02-09; First posted 2019-02-15 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Spinal Deformity; Trauma; Spinal Tumor; Surgical Site Infection
Keywords: vancomycin powder; surgical site infection; open posterior spinal surgery
MeSH Terms: conditions — Wounds and Injuries; Spinal Cord Neoplasms; Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: Single-blinded open-label randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: This will be a single blinded trial as patients will not know their treatment allocation until the termination of study. Operating surgeons cannot be blinded to allocation. However, all clinical and radiological outcomes will be evaluated by an independent researcher who is blinded to the allocation. This researcher will be blinded to the study treatment throughout the study period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Vancomycin (Active Comparator): Intervention: 1g vancomycin powder locally applied to the deep wound and subcutaneous layer prior to closure.
  Interventions: Drug: Vancomycin powder
- Control - No vancomycin application (No Intervention): No intervention, control group All other wound closure procedure and wound care and monitoring are the same

INTERVENTIONS:
Drug: Vancomycin powder — For the intervention group, the use of 1g vancomycin powder to be placed in the deep wound and subcutaneous layer prior to closure.
  Arms: Intervention - Vancomycin

SUMMARY:
Surgical site infections (SSI) are not uncommon, especially in specific high-risk groups including spinal deformity and tumor (i.e. metastatic spine surgery) surgery. Well-recognized measures have been adopted to reduce surgical site infection, and the use of topical vancomycin powder has gained popularity in recent years. Given the lack of high-quality evidence for the use of topical vancomycin to reduce surgical site infections in open posterior spine surgery, which is currently the most common approach to spine surgery, it is crucial to study the use of vancomycin powder in reducing surgical site infections. This study is a prospective, single-blinded open label randomized controlled trial, with one arm of patients having local administration of 1g vancomycin powder which will be placed in the deep wound and subcutaneous layer prior to closure of surgical site by the orthopaedic surgeon, whereas the control arm will be without such application of vancomycin. Both arms of patients will still be undergoing the same operation procedures, as well as postoperative local wound drainage and wound care. This study will provide insights on the reduction rate in superficial and/or deep surgical site infection, and also assess the cost-effectiveness of using topical vancomycin in reducing surgical site infection between different disease groups, as well as any postoperative serum vancomycin toxicity and renal impairment. These proposed findings will provide valuable information for clinicians and institutions on future measures for surgical site infection of open posterior spine surgery.

DETAILED DESCRIPTION:
Objectives:

Primary Objectives:

To evaluate the efficacy of intra-wound administration of vancomycin powder as add-on prophylactic intraoperative antibiotic in patients at high risk for surgical site infections after receiving open posterior spinal surgery

Secondary Objectives:

* To evaluate the safety of intra-wound administration of vancomycin powder as an add-on prophylactic intraoperative antibiotic
* To evaluate the cost-effectiveness of intra-wound administration of vancomycin powder as an add-on prophylactic intraoperative antibiotic compared to standard prophylactic intraoperative care

Hypothesis to be tested:

The intra-wound vancomycin powder as add-on prophylactic intraoperative antibiotic can significantly reduce the rate of surgical site infection.

Design and subjects:

The study is a prospective, parallel group, single-blinded randomized controlled trial.

All eligible patients who have consented to take part in the study will be randomized to either intervention or control group with a 1:1 allocation ratio. Patients allocated to the intervention group will receive intra-wound vancomycin powder 1gram as add-on prophylactic intraoperative antibiotic during the surgery. Patients allocated to the control group will not receive any add-on prophylactic intraoperative antibiotic. Patients will not know their treatment allocation until study termination.

Surgical site condition of all the patients will be assessed after the surgery. Investigator will examine the surgical wound and observe any signs and/or symptoms of SSI during hospitalization and follow-up visits until 1 year post-operation. For patients received instrumentation and fusion operation, additional radiographs of the operated sites will be performed for assessing any implant loosening and non-union at 3, 6 and 12 months postoperatively. All clinical and radiological outcomes will be evaluated throughout the study period.

Instruments: Parameters include age, gender, smoking and drinking history, pathology (deformity, tumor, trauma, degenerative), location and spinal levels of surgery, if instrumentation is used, operative time, blood loss, need for transfusion, significant co-morbidities including diabetes mellitus, renal failure, immunocompromised state, and dural tear events.

Interventions: Patients are randomized into the treatment group where 1g of vancomycin powder is administered to the deep and superficial spinal wound, and the control group without vancomycin powder use.

Main outcome measures: Primary outcome is the rate of surgical site infection. Secondary outcomes include vancomycin toxicity measured by vancomycin levels and renal function for three consecutive postoperative days, and cost-effectiveness calculation for each disease group. Additionally for those undergoing fusion surgery, 1-year follow-up assessment for fusion rates.

Data analysis:

For descriptive statistics, means and standard deviations or medians and interquartile ranges will be presented for continuous variables, frequencies and percentages will be presented for categorical/ discrete variables.

Baseline Comparison The baseline characteristics of the intervention and control group will be evaluated. The Student's t-test or Wilcoxon Rank-Sum test (according to the frequency distribution of the variables studied) will be used to compare continuous variables, and Chi-square or Fisher's exact test will be used to compare categorical/discrete variables.

Primary Efficacy Analysis Fisher's exact test will be performed to evaluate the difference of SSI rates between the intervention and control group. The respective 95% confidence interval (CI) will be calculated and presented. If it is appropriate, the adjustment for baseline covariates will be made to the primary efficacy comparison. The analysis will primarily be carried out according to ITT population and subordinately based on PP population. Both ITT and PP results will be reported.

Adjusted Analysis for Confounding Factors:

If baseline imbalance is observed, adjustment for confounding factors in the primary analysis will be investigated by a multiple logistic regression for the potential risk factors with SSI as follows:

* Patient-related risk factors include socio-demographics and co-morbidities including, diabetes mellitus, ischemic heart disease, chronic obstructive pulmonary disease, renal impairment/failure, immunocompromised state and nutritional deficiency.
* Procedure-related risk factors include type and site of surgery, intraoperative details including number of spinal level operated, length of instrumentation, use of fusion, use of drain, operation duration, presence of dural tear and number of surgeons in operating room
* Intra- and post-operative blood loss and blood product transfusion.

Cost-effectiveness analysis The cost-effectiveness analysis will estimate the Incremental cost-effectiveness ratio(ICER), which is the incremental cost per SSI prevented for the add-on administration of vancomycin powder compared with standard care over a 1-year post-operative period.

The total cost for SSI will be calculated by multiplying the quantity of resource use by unit costs. Future costs will be discounted at a rate of 3% per year.

Non-parametric bootstrapping will be used to determine the 95% CIs for ICERs. A non-parametric bootstrap replications of 1000 with replacement generating multiple data sets from the original data will be used. In each dataset, the statistic of interest (mean costs, SSIs, and ICERs) will be calculated. Multiple sensitivity analysis will be performed to evaluate the robustness of the findings.

Uncertainty in the estimates of the cost-effectiveness evaluation will be visualized by plotting the cost-effectiveness plane and acceptability curves. The acceptability curves will be used to determine the probability that the additional use of vancomycin powder will be cost-effective compared with standard care, at different values of ceiling ratio or acceptable willingness-to-pay threshold.

The cost-effectiveness analysis will be carried out according to the ITT population.

Safety Analysis The incidence of adverse effects (AEs) will be summarized by system organ class and severity grading according to the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Event (CTCAE) version 5. AEs will be tabulated by severity grading and relationship with study intervention.

The AESIs will be summarized in similar manner as all AEs. The safety analysis will be carried out according to in the safety population.

Expected results: Intra-wound administration of vancomycin powder reduces surgical site infections, is not toxic, and the most cost-effective disease groups are deformity correction and tumor surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male adult with age ≥18 years
2. Undergoing open posterior spinal surgery with instrumentation indicated for spinal deformity, trauma and tumor
3. Able to understand the nature, scope and possible consequences of participation in the study
4. Appropriate voluntary written informed consent have been provided by patients

Exclusion Criteria:

1. Has been treated with antibiotics due to primary spinal infection (i.e. spondylodiscitis) within 1 year prior to surgery
2. Ongoing treatment with antibiotics for other infections
3. Undergoing minimally invasive surgery or anterior-only surgical approaches or deformity correction surgery for adolescent idiopathic scoliosis (inherent low-risk for surgical site infections18)
4. Undergoing decompression-only surgery for cervical spine, spinal deformity, trauma and tumors
5. Has known history of allergy to vancomycin, penicillin and other glycopeptides (teicoplanin)
6. Has history of vancomycin resistance
7. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of superficial incisional SSI | one year
  CDC Surgical Site Infection Criteria (Centers for Disease Control, Procedure-associated Module SSI, January 2019)
  The definition of SSSI is:
  1. an infection occurs within 30 days after operation (where day 1= operation day);
     AND
  2. Involves only skin/subcutaneous tissue of the incision;
  AND
  3) Patient has at least one of the following: a)purulent drainage from the superficial incision; b)organism(s) identified from an aseptically-obtained specimen from the superficial incision or subcutaneous tissue by a culture/non-culture based microbiologic testing method; c)superficial incision being deliberately opened by a surgeon, attending doctor/other designee and culture/non-culture based testing of the superficial incision or subcutaneous tissue is not performed AND Patient has at least one of the following: localized pain/tenderness, localized swelling, erythema, or heat; d) SSSI diagnosed by a surgeon, attending doctor/other designee.
Incidence of deep incisional SSI | one year
  Deep Incisional SSI (DSSI)
  1. For deep incisional SSI, the definition is an infection occurring within 90 days after the operation (where day 1 = the procedure day); AND
  2. Involves deep soft tissues of the incision (e.g. fascial and muscle layers); AND
  3. Patient has at least one of the following:
     1. purulent drainage from the deep incision;
     2. a deep incision spontaneously dehisces, or is deliberately opened or aspirated by the surgeon, attending doctor or other designee;
        AND
        Organism(s) identified from the deep soft tissues of the incision by a culture or non-culture based microbiologic testing method which is performed for purposes of clinical diagnosis or treatment;
        AND
        Patient has at least one of the following signs and symptoms: fever (>38 °C); localized pain or tenderness;
     3. An abscess or other evidence of infection involving the deep incision that is detected on gross anatomical or histopathologic exam, or imaging test.
Number of participants with adverse event (AE) to vancomycin | one year
  An AE is any untoward medical occurrence to a patient which does not necessarily has a causal relationship with the study intervention, and it can also occur outside of the time period. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), new or exacerbated symptoms/diseases temporally associated with the study intervention, whether or not the event is considered causally related to the use of intervention. Medical conditions/diseases present before the study intervention are only considered as AEs if they worsen after intervention. Signs and symptoms that are clearly due to natural process of underlying disease/disease progression should not be reported. SSSI/DSSI is not regarded as an AE in the study. Secondary infection of a SSSI/DSSI or other infection shall be regarded as an AE.
  The term AE is used to include both serious and non-serious AE.

SECONDARY OUTCOMES:
Cost-effectiveness of vancomycin use | one year
  Determination of which disease group is most cost-effective in terms of cost per surgical site infection episode reduced. Will identify the highest risk group (i.e. deformity or tumor surgery) and see whether the risk of infection is significantly different between intervention and control groups as compared to perceived less risk groups (i.e. simple decompression surgery, no implants). Cost items include cost of vancomycin drug, hospitalization days, prolonged antibiotic use, repeated operations for debridement
Incremental cost-effectiveness ratio | one year
  It is the incremental cost divided by the difference in the number of SSI cases between treatment group and control group over a 1-year post-operative period.
Serum vancomycin level | Three days postoperatively
  3 days postoperative serum assessment of vancomycin levels to identify any vancomycin toxicity in serum
Renal function test | Three days postoperatively
  3 days postoperative serum assessment of renal function tests to identify any renal impairment

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No